CLINICAL TRIAL: NCT04356755
Title: Subcutaneous Injections of Cultured Adipose-derived Stroma/ Stem Cells to Heal Refractory Ischemic Digital Ulcers in Patients With Scleroderma
Brief Title: Subcutaneous Injections of ASC to Heal Digital Ulcers in Patients With Scleroderma.
Acronym: ADUSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/17/0447
Record Dates: First submitted 2020-03-11; First posted 2020-04-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AdMSC (Experimental): Subcutaneous injections of cultured adipose-derived stroma/stem cells to heal refractory ischemic digital ulcers in patients with scleroderma
  Interventions: Drug: AdMSC
- Placebo (Placebo Comparator): Subcutaneous injections of placebo comparator to heal refractory ischemic digital ulcers in patients with scleroderma
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AdMSC — At day 0, patients will have AdMSC injections in their ischemic DU. Patients will be followed-up for 16 weeks
  Arms: AdMSC
Drug: Placebo — At day 0, patients will have placebo injections in their ischemic DU. Patients will be followed-up for 16 weeks
  Arms: Placebo

SUMMARY:
Ischemic digital ulcers (DUs) are a frequent complication in systemic sclerosis with a major impact on hand function and quality of life. Digital injection of cultured adipose-derived stromal cell (AdMSC) constitutes a promising approach to treat scleroderma-induced refractory ischemic DUs where no alternative therapy is validated. The aim of this phase 2 study is to compare efficacy and safety of digital injection of AdMSC versus placebo for healing refractory active ischemic digital ulcers in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a systemic autoimmune disease characterized by an autoimmune-mediated microangiopathy and progressive fibrosis. Ischemic digital ulcers (DUs) are frequent in the disease course. DUs are an expression of the severity of the microangiopathy. DUs lead to pain, infection, gangrene, autoamputation, impaired hand use and impaired quality of life. The management of DUs is often based on optimal wound care to promote healing and and repeated hospitalizations to perform onerous prostacyclin infusions to reduce pain and accelerate healing. With optimal standard of care, only 60% of DUs are healed after 3 months and 46.2% experiences recurrence during that time among them 11.2% experiences a chronic evolution. No drug has demonstrated a positive effect on refractory DUs healing. The rational underlying the use of cultured adipose-derived stromal cell (AdMSC) in this indication is based on the finding of AdMSC, in vitro and in vivo, angiogenic and anti-inflammatory potential in other ischemic pathologies, with an excellent safety profile. The pilot phase of the ACellDREAM trial demonstrated the feasibility and safety of AdMSC transplantation in patients with non- revascularizable critical limb ischemia and showed improvement in ulcer evolution and wound healing. The EFS-O culture procedure safety is validated and is already in use in ongoing French and European clinical trials. Two pilot studies showed the safety of adipose tissue grafting for scleroderma-Induced DU. The SCLERADEC pilot study outlines the safety, in 12 SSc patients, of the digital injection of adipose- derived stromal vascular fraction, which is a heterogeneous population of cells including only 36% of uncultured AdMSC. An improvement in hand disability, quality of life and DUs was observed, the phase II is ongoing. The hypothesis of the study is that digital injection of AdMSC could be efficacious for scleroderma-induced refractory ischemic DUs healing by digital vascular regeneration in a clinical situation where no alternative therapy is validated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years of age,
* Patient with systemic sclerosis according to the 2013 ACR/EULAR classification criteria9,
* SSc patient with at least one refractory active ischemic digital ulcer at "inclusion visit" (see below the eligibility conditions of a DU),
* Age > 50 years and not treated with any kind of hormone replacement therapy for at least 2 years prior to screening, with amenorrhea for at least 24 consecutive months prior to screening. An assessment of serum follicle stimulating hormone showing a level of > 40 TU/L at screening may be used to exclude childbearing potential, based on the discretion of the investigator,
* Patient must have provided written informed consent prior to enrolment,
* Patient must be able to understand their requirements of participating in the protocol,
* Patient affiliated to a social security system.
* Relative to each DU :

The DU at " inclusion visit " must show all the following characteristics:

1. Located beyond the proximal interphalangeal joint, on finger surface (included periungual ulcers),
2. Of ischemic origin according to the physician,
3. Not over subcutaneous calcifications or bone relief,
4. Active DU,
5. Refractory after 10±2 weeks of standard of care according to EULAR recommendations26 (that is either still active (chronic) or new occurrence despite standard of care)

Exclusion Criteria:

* Current smoker or tobacco consumption stopped for less than 3 months prior to inclusion, - Patient participating in a clinical trial or having participated in a clinical trial within the previous 3 months,
* Patients on statins, who have received treatment for less than 3 months prior to Screening or whose treatment has not been stable during this period,
* Patients on vasodilators, such as endothelin receptor antagonists (ERAs), PDE5 inhibitors (e.g. sildenafil, tadalafil), calcium channel blockers, ACE-inhibitors, nitroglycerin, alpha adrenergic blockers, or angiotensin II receptor antagonists, N-acetylcysteine, antiplatelet aggregation therapy and low molecular weight heparin who have received treatment if present for less than 3 months prior to "inclusion visit" or whose treatment has not been stable for at least 1 month prior to "inclusion visit",
* Treatment with disease modifying agents such as methotrexate, mycophenolate mofetil, azathioprine, tacrolimus, Interferons and cyclophosphamide, those drugs should be stop at least 1 month prior study entry.
* Treatment with oral corticosteroids (> 10 mg/day of prednisone or equivalent),
* Systemic antibiotics (oral and TV) to treat infected DU(s) within 4 weeks prior to "inclusion visit",
* Use of topical growth factors, hyperbaric oxygen,
* Local injection of botulinum toxin in an affected finger within 4 weeks prior to "inclusion visit",
* Surgical sympathectomy of the upper limbs or surgical wound debridement within 1 month prior to "inclusion visit",
* Liposuction technically impossible,
* Patient who underwent autologous hematopoietic stem cell transplantation (HSCT) within less than 1 year,
* Patients with an indication for intensification by autologous HSCT (according to EBMT guidelines and national RCP MATHEC),
* History of cancer in the last five years, except for successfully excised basal cell/squamous cell carcinoma, or successfully excised early melanoma of the skin. Subjects, who had successfully tumor resection or radiation or chemotherapy more than 5 years from inclusion and no recurrence, may be enrolled in the study, - Subjects who have active proliferative retinopathy,
* Positive HIV-1 or 2, HTLV-1 or 2, HBV or HCV,
* Patients with a history of stroke, myocardial infarction or severe arrhythmia in the last 6 months
* Patient who had severe cardiac failure in the last 6 months,
* Females who are pregnant or breastfeeding or plan to do so during the course of this study,
* Patient under judicial protection, - Refusal of the patient to participate in the study.
* Relative to each DU:

  1. Digital ulcer due to conditions other than scleroderma,
  2. Non ischemic digital ulcer,
  3. Ulcers with osteomyelitis, or clinically uncontrolled infection,
  4. Infected digital ulcer requiring systemic antibiotherapy,
  5. Digital ulcer requiring urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of refractory active ischemic digital ulcers healed (complete or partial) | 16 weeks
  Partial healing is defined as > 50% reduction of the DU area or > 50% re epidermisation of the DU.
Composite endpoint combining healing (complete or partial) without recurrence and without local or general complications | 16 weeks
  Partial healing is defined as > 50% reduction of the DU area or > 50% re epidermisation of the DU.
  Local complications resulting from DU worsening:
  * Critical ischemic crisis necessitating hospitalization,
  * Gangrene, (auto) amputation,
  * Failure of conservative management: Surgical and chemical sympathectomy, vascular reconstructions, or any unplanned surgery in the management of hand SSc manifestation(s),
  * Use of parenteral prostanoids after treatment injection,
  * Requiring class II, III or IV narcotics or increase in existing dose of > 50 % as compared to baseline,
  * Initiation of systemic antibiotics for the treatment of infection attributed to digital ulceration.
  General complications will be assessed by:
  * Clinical examination
  * Patient reported-outcomes
  * Laboratory assessments

SECONDARY OUTCOMES:
Percentage of participants with Digital Ulcer complete healing | 16 weeks
  Number of complete ulcer Healing. Complete healing is defined as 100% re-epidermisation.
Percentage of participants with Digital Ulcer partial healing | 16 weeks
  Number of partial ulcer Healing. Partial healing is defined as > 50% reduction of the DU area or > 50% re epidermisation of the DU.
Percentage of participants with wound surface reduction <50% | 16 weeks
  the wound surface reduction is defined by analysis photography
Percentage of participants with new Digital Ulcer | 16 weeks
  Number of patients who do not develop any new DU.
Percentage of participants with Digital Ulcer complication | 16 weeks
  A complication is an infection, gangrene, amputation or a DU requiring IV prostanoids.
Change from Baseline in Pain Scores | 16 weeks
  Evaluation of pain on a Visual Analog Scale. The visual scale measures the intensity of pain on a scale ranging from 0 (no pain) to 10 (maximum pain).
Change from Baseline in severity of Raynaud's phenomenon | 16 weeks
  Change in severity of Raynaud's phenomenon on a Visual Analog Scale. The visual scale is in a form of plastic ruler and measures the severity of Raynaud's phenomenon on a scale ranging from 0 (no pain) to 100 (maximum pain).
Change from Baseline in Digital ischaemia | 16 weeks
  Change in digital ischaemia of the treated fingers on Digital arterial pressure.
Change from Baseline in cutaneous ischaemia | 16 weeks
  Change in cutaneous ischaemia of the treated fingers on transcutaneous oxygen pressure (TcPO2).
Change from Baseline in Digital microvascular organisation | 16 weeks
  Change in digital microvascular organisation of the treated fingers on nailfold capillaroscopy.
Change from Baseline in hand functional disability | 16 weeks
  Evaluation of hand functional disability by the Cochin Hand Function Scale.
Change from Baseline in quality of life in systemic sclerosis | 16 weeks
  Evaluation of quality of life in systemic sclerosis by scleroderma health assesment (SHAQ).
Change from Baseline in quality of life | 16 weeks
  Evaluation of quality of life by the SF36.
Change from Baseline in health status | 16 weeks
  Evaluation of health status by the EQ5D.
Vascular biomarkers | 16 weeks
  Endothelin-1, Endostatin, Endogline, Angiotensin I and II, Tie 1 and 2, V-EGF, sICAM-1, sVCAM, E-selectin, CXCL4 plus anti-AT1R, anti-ETAR, anti Annexin V will be measured out in blood samples by Luminex

CONTACTS AND LOCATIONS:
Overall Officials: Grégory PUGNET, MD, PHD, Principal Investigator
Locations (7):
- France (7):
  - Grenoble Hospital, Grenoble
  - Lille Hopsital, Lille
  - Marseille Hospital, Marseille
  - Montpellier Hospital, Montpellier
  - Nantes Hospital, Nantes
  - Poitiers Hospital, Poitiers
  - CHU de Toulouse - Hôpital PURPAN-TSA, Toulouse